CLINICAL TRIAL: NCT06852495
Title: A Study of Colorectal Cancer Development and Prognosis Based on Environmental Factors and Macrogenomes
Brief Title: the Effect of Environmental Factors on Colorectal Cancer Based on Macrogenomes
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-443-01
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Colorectal cancer; Macrogenome; Environmental pollution; air pollution
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the colorectal cancer group: patients diagnosed with colorectal cancer
- the control group: Healthy individuals with no history of malignant tumor

SUMMARY:
The aim of this study is to investigate the effects of environmental factors, such as air pollution, on the occurrence, development and prognosis of colorectal cancer; to identify metabolic markers specific to colorectal cancer patients, which will provide a basis for early diagnosis, early intervention and individualized treatment; and to comprehensively understand the mechanism of the occurrence and development of colorectal cancer by integrating the data of environmental factors and the macro-genome, and to develop new predictive and therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Patients diagnosed with colorectal cancer by pathologic biopsy before surgery;
* Patients did not undergo chemotherapy, radiotherapy, targeted and immunotherapy, etc. before enrollment;
* Willing to participate in the study and sign an informed consent form. Complete clinical data.

Exclusion Criteria:

* Concurrent primary malignant tumor other than colorectal cancer;
* Patients with severe cardiopulmonary insufficiency or other systemic diseases that affect the choice of treatment plan;
* Inappropriate for enrollment as assessed by the investigator;
* Incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with colorectal cancer by pathological biopsy and healthy participants with no history of malignancy were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
prognosis | From date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first, assessed up to 60 months
  Overall survival (OS), from date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first.

SECONDARY OUTCOMES:
Macrogenomic differences | The date of macrogenomic testing, assessed up to 1 week after surgery.
  Macrogenomic differences in feces.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data sharing is not permitted by the Ethics Committee of the First Affiliated Hospital of Chongqing Medical University.